CLINICAL TRIAL: NCT04262076
Title: Effect of Pulpine and Combination of Pulpine With Polyamidoamine Dendrimer on Remineralization of Carious Affected Human Dentin
Brief Title: Remineralization of Caries Affected Dentin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mona Rizk Abo El Wafa Ahmed, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC17-01123
Record Dates: First submitted 2020-01-26; First posted 2020-02-10 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Deep Caries

STUDY DESIGN:
Intervention Model Description: split mouth design
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of pulpine with Polyamidoamine Dendrimer (Experimental): Removal of Caries infected dentin from the walls and floor of the cavity and then apply polyamidoamine Denrimer for 30 secs ,then washed out of the cavity followed by placement of Pulpine over affected Dentin.
  Interventions: Other: Pulpine with Polyamidoamine Dendrimer
- Pulpine (Active Comparator): Removal of Caries infected dentin from the walls and the floor of the cavity followed by application of Pulpine over affected Dentin.
  Interventions: Other: Pulpine with Polyamidoamine Dendrimer

INTERVENTIONS:
Other: Pulpine with Polyamidoamine Dendrimer — Removal of infected dentin in class I Cavities followed by application of Polyamidoamine Denrimer on caries affected Dentin that is washed out of the cavity after 30 secs then finally place Pulpine .

SUMMARY:
Remineralization of carious affected dentin

DETAILED DESCRIPTION:
Remineralization of Carious affected dentin by using Pulpine alone and combination of Pulpine with Polyamidoamine Dendrimer.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one class one carious posterior teeth in both left and right side.
* Absence of spontaneous pain, Mobility and tenderness on percussion.
* Radiographically, the preoperative inclusion criteria are, no internal or external resorption and no widening of the periodontal membrane space.

Exclusion Criteria:

* Patients with poor oral Hygiene.
* Evidence of Rampant Caries.
* Teeth with periodontal involvement.
* Poor general health condition.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Remineralization & increase dentin density that is measured by using Vista Scan Radiography. | 6 months
  Vista scan Radiography used to measure pixel grey value after 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Faculty of Dentistry for Girls, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol